CLINICAL TRIAL: NCT06626958
Title: The Effect of the Stress Ball Used in the Active Phase of Labor on Labor Pain and Birth Comfort
Brief Title: Stress Ball Used in the Active Phase of Labor on Labor Pain and Birth Comfort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sibel ÖZTÜRK, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SOZTURK0004
Record Dates: First submitted 2024-09-18; First posted 2024-10-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Labor Pain; Birth Order; Stress
Keywords: Active phase of labor,; stress ball,; labor pain,; labor comfort
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental trial
Who Masked: Outcomes Assessor
Masking Description: The researcher performing the statistical analysis will not know which data is the experimental group and which is the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vsisual Analog Scale (VAS) (Experimental): The VAS scale will be used to evaluate the level of labor pain in the intervention and control groups.
  Interventions: Behavioral: Stress Ball
- Labor Comfort Scale (Experimental): The birth comfort scale will evaluate the birth comfort of women in the intervention and control groups during birth.
  Interventions: Behavioral: Stress Ball

INTERVENTIONS:
Behavioral: Stress Ball — Stress Ball app

SUMMARY:
The aim of the clinical trial is to examine the effect of a stress ball applied to pregnant women during the active phase of labor on labor pain and labor comfort. The effect of the stress ball used in the experimental group on labor pain and labor comfort will be evaluated. The stress ball applied to pregnant women during the active phase of labor minimizes labor pain and increases labor comfort H 0: The stress ball used during the active phase of labor has no effect on labor pain and labor comfort.

H 1: The stress ball used during the active phase of labor increases labor pain and labor comfort.

The researchers will monitor the pregnant women from the time the cervical dilation is 3-4 cm (from the active phase of labor) until the cervical dilation is 8-9 cm and the experimental group will be asked to use the stress ball. Routine application will be made to the control group. The pain during labor of the experimental and control groups will be evaluated with the VAS scale. After the birth, the labor comfort scale will be applied to measure labor comfort.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal birth
* Pregnant women between the ages of 18-40

Exclusion Criteria:

* Risky pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Labor pain and labor comfort will be evaluated.
Enrollment: 140 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-03-26 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Lapor Pain | First measurement: Within the first hour of labor Second Measurement: Within 10-12 hours of labor
  The VAS scale will be used to evaluate the level of labor pain in the intervention and control groups. VAS is scored from 1 to 10. As the score obtained from the scale increases, it shows that the labor pain also increases. After the pre-test and the intervention, it is expected that the pain will change in the interventionl group and the VAS score will change.Measurement will begin when cervical dilation is 3-4 cm, and the final test will be performed and completed when cervical dilation is approximately 7-8 cm. This will take approximately 10-12 hours.
Labor Comfort | First measurement: Within the first hour of labor Second Measurement: Within 10-12 hours of labor
  The minimum score on the scale is 9 and the maximum score is 45. It indicates that as the score value of the scale increases, comfort increases, and as the score value decreases, comfort decreases.The minimum score on the scale is 9 and the maximum score is 45. As the score of the scale increases, it indicates that comfort increases, and as the score decreases, comfort decreases. The birth comfort scale will be applied when the cervical dilatation reaches 7-8 cm. It is expected that the birth comfort will be higher in the intervention group than in the experimental group. The scale will be applied within the first hour when the cervical dilatation reaches 7-8 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Mihriban Elmas, Principal Investigator — mihriban.elmas@icloud.com
Locations (1):
- Muş State Hospital Birth Hall, Muş, Merkez, Turkey (Türkiye)